CLINICAL TRIAL: NCT00289224
Title: A Randomized Controlled Trial of the Bivalent Killed Whole Cell Oral Cholera Vaccine in Eastern Kolkata, West Bengal, India
Brief Title: Randomized Controlled Trial of Killed Oral Cholera Vaccine in Kolkata
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: International Vaccine Institute (Other)
Collaborators: National Institute of Cholera and Enteric Diseases, India (Other); Shantha Biotechnics Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C8phIII
Record Dates: First submitted 2006-02-07; First posted 2006-02-09 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2012-03

CONDITIONS: Diarrhea; Cholera; Vibrio Infections
Keywords: bivalent killed whole cell oral cholera vaccine; double blind randomized clinical trial
MeSH Terms: conditions — Diarrhea; Cholera; Vibrio Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Cholera Vaccine
  Interventions: Biological: bivalent killed whole cell oral cholera vaccine
- 2 (Placebo Comparator): Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: bivalent killed whole cell oral cholera vaccine — Given as 1.5 mL dose, given orally in 2 doses 14 days apart, each dose contains:
  V. cholerae O1 Inaba El Tor strain Phil 6973 formalin killed 600 Elisa units (EU) LPS V. cholerae O1 Ogawa classical strain Cairo 50 heat killed 300 EU LPS V. cholerae O1 Ogawa classical strain Cairo 50 formalin killed 300 EU LPS V. cholerae O1 Inaba classical strain Cairo 48 heat killed 300 EU LPS V. cholerae O139 strain 4260B formalin killed 600 EU LPS
  Arms: 1
Biological: Placebo — Heat Killed E. coli K12 in an optical turbidity identical to killed oral cholera vaccine, in 1.5 mL oral dose given twice, at least 14 days apart.
  Arms: 2

SUMMARY:
The primary purpose of this study is to estimate the efficacy of a two-dose regimen of the oral killed bivalent cholera vaccine when administered to individual residing in a cholera-endemic area in India.

DETAILED DESCRIPTION:
Cholera remains a serious public health problem worldwide. Provision of safe water and food, establishment of adequate sanitation, and implementation of personal and community hygiene constitute the main public health interventions against cholera. These measures cannot be implemented fully in the near future in most cholera-endemic areas. A safe, effective, and affordable vaccine would be a useful tool for cholera prevention and control.The World Health Organization recently recommended that the newer generation cholera vaccines be considered in certain endemic and epidemic situations, but indicated that demonstration projects are needed to provide more information about the costs, feasibility, and impact of using these vaccines. Starting in the mid-1980s, following technology transfer from Prof Jan Holmgren in Sweden, Vietnamese scientists at the National Institute of Hygiene and Epidemiology (NIHE) in Hanoi developed and produced an oral, killed cholera vaccine for the country's public health programs (10). Since licensure of the oral cholera vaccine in Vietnam, more than 5 million doses have been administered without any report of serious adverse events.

The vaccine is produced according to recommended WHO guidelines (6) at the NIHE's newly privatized arm, the Company for Vaccine and Biological Production No. 1 (VABIOTECH) in Hanoi. Recently the vaccine was reformulated in order to comply with WHO standards to further internationalize this vaccine. Phase II trials of this reformulated vaccine have been performed among 148 adults in SonLa,Vietnam (18) and among 100 adults and 100 children in Kolkata, India. Results from these trials reveal that the vaccine is safe and immunogenic.

A double-blind randomised phase III trial of the reformulated oral killed bivalent cholera vaccine in an urban slum site in Kolkata is proposed by the National Institute of Cholera and Enteric Diseases (NICED) in collaboration with the International Vaccine Institute (IVI). The IVI has negotiated an agreement between VABIOTECH and Shantha Biotechnics PVT LTD for the vaccine and placebo to be used during the trial. VABIOTECH will produce bulk oral killed bivalent cholera vaccine under quality control conditions to be supervised by IVI staff. Shanta will purchase bulk vaccine from VABIOTECH, fill and finish the bulk vaccine, and obtain regulatory clearance for use of the vaccine in the phase III trial. Shanta will purchase the bulk placebo agent for use in the trial from IVAC (also in Vietnam) and Shanta will fill and finish the placebo and obtain regulatory clearance for use of the placebo in the phase III trial. Shanta will later obtain the technology for future production of the oral killed bivalent cholera vaccine. The results of this trial will pave the way for the use of this vaccine in India and other cholera-endemic areas.

ELIGIBILITY:
Inclusion Criteria:

* All healthy, consenting, non-pregnant (as ascertained by history) residents at least 1 year of age of the study area

Exclusion Criteria:

* individuals who are too weak to get out of bed to receive the vaccine;
* pregnant women (identified through verbal screening); and
* those less than 1 year of age

Min Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 69329 (Actual)
Dates: Start 2006-07; Primary Completion 2011-12 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
culture-proven V. cholerae O1 diarrhoea episodes severe enough to require treatment in a health care facility. | 1095 days

SECONDARY OUTCOMES:
Episodes of acute watery diarrhoea severe enough to require treatment in a health care facility | 1095 days
Serum vibriocidal responses, compared to baseline | 14 days and 365 days after second dose

CONTACTS AND LOCATIONS:
Overall Officials: Dipika Sur, MD, Principal Investigator — National Institute of Cholera and Enteric Diseases, India
Locations (1):
- National Institute of Cholera and Enteric Diseases, Kolkata, West Bengal, India

REFERENCES:
- [Result] Sur D, Lopez AL, Kanungo S, Paisley A, Manna B, Ali M, Niyogi SK, Park JK, Sarkar B, Puri MK, Kim DR, Deen JL, Holmgren J, Carbis R, Rao R, Nguyen TV, Donner A, Ganguly NK, Nair GB, Bhattacharya SK, Clemens JD. Efficacy and safety of a modified killed-whole-cell oral cholera vaccine in India: an interim analysis of a cluster-randomised, double-blind, placebo-controlled trial. Lancet. 2009 Nov 14;374(9702):1694-702. doi: 10.1016/S0140-6736(09)61297-6. Epub 2009 Oct 8. PMID 19819004
- [Derived] Islam MT, Im J, Ahmmed F, Kim DR, Tadesse BT, Kang S, Khanam F, Chowdhury F, Ahmed T, Firoj MG, Aziz AB, Hoque M, Park J, Jeon HJ, Kanungo S, Dutta S, Zaman K, Khan AI, Marks F, Kim JH, Qadri F, Clemens JD. Better Existing Water, Sanitation, and Hygiene Can Reduce the Risk of Cholera in an Endemic Setting: Results From a Prospective Cohort Study From Kolkata, India. Open Forum Infect Dis. 2023 Nov 21;10(11):ofad535. doi: 10.1093/ofid/ofad535. eCollection 2023 Nov. PMID 38023545
- [Derived] Fong Y, Halloran ME, Park JK, Marks F, Clemens JD, Chao DL. Efficacy of a bivalent killed whole-cell cholera vaccine over five years: a re-analysis of a cluster-randomized trial. BMC Infect Dis. 2018 Feb 20;18(1):84. doi: 10.1186/s12879-018-2981-4. PMID 29463233
- [Derived] Ali M, Debes AK, Luquero FJ, Kim DR, Park JY, Digilio L, Manna B, Kanungo S, Dutta S, Sur D, Bhattacharya SK, Sack DA. Potential for Controlling Cholera Using a Ring Vaccination Strategy: Re-analysis of Data from a Cluster-Randomized Clinical Trial. PLoS Med. 2016 Sep 13;13(9):e1002120. doi: 10.1371/journal.pmed.1002120. eCollection 2016 Sep. PMID 27622507
- [Derived] Ali M, Sur D, You YA, Kanungo S, Sah B, Manna B, Puri M, Wierzba TF, Donner A, Nair GB, Bhattacharya SK, Dhingra MS, Deen JL, Lopez AL, Clemens J. Herd protection by a bivalent killed whole-cell oral cholera vaccine in the slums of Kolkata, India. Clin Infect Dis. 2013 Apr;56(8):1123-31. doi: 10.1093/cid/cit009. Epub 2013 Jan 29. PMID 23362293
- [Derived] Sur D, Kanungo S, Sah B, Manna B, Ali M, Paisley AM, Niyogi SK, Park JK, Sarkar B, Puri MK, Kim DR, Deen JL, Holmgren J, Carbis R, Rao R, Nguyen TV, Han SH, Attridge S, Donner A, Ganguly NK, Bhattacharya SK, Nair GB, Clemens JD, Lopez AL. Efficacy of a low-cost, inactivated whole-cell oral cholera vaccine: results from 3 years of follow-up of a randomized, controlled trial. PLoS Negl Trop Dis. 2011 Oct;5(10):e1289. doi: 10.1371/journal.pntd.0001289. Epub 2011 Oct 18. PMID 22028938